CLINICAL TRIAL: NCT06687317
Title: Reliabılıty,Validity Of The Turkish Version Of The KNAP
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, GÖKHAN MARAŞ, Research assistant, Amasya University
Other Study IDs: 2024-11
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Other
Keywords: Validity; Reliability; Version
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Behavioral — KNAP
  Other Names: Observational

SUMMARY:
This study, we performed the Turkish version validity and reliability of the KNAP

DETAILED DESCRIPTION:
Chronic musculoskeletal pain is significantly affected by the attitudes and beliefs of healthcare professionals and affects patient management outcomes . Adopting a biopsychosocial approach rather than a solely biomedical approach is of great importance in order to comply with current pain management guidelines and reduce both pain levels and disability . Therefore, it is important to recognize healthcare professionals' knowledge, attitudes, and beliefs regarding pain . Pain science education is a powerful strategy to manage chronic musculoskeletal pain by addressing biopsychosocial factors . It improves the understanding of pain by integrating psychological and social aspects beyond anatomical factors and provides better rehabilitation outcomes. Healthcare professionals are crucial to providing effective treatment and patient pain education and require a solid understanding of pain science principles . Many validated surveys assess health care professionals' knowledge and attitudes regarding chronic pain, but they often lack elements of modern pain science and biopsychosocial treatment orientations . To address these limitations, the Knowledge and Attitudes to Pain (KNAP) questionnaire was developed to assess modern pain science and biopsychosocial attitudes toward pain. The KNAP questionnaire consists of 30 items divided into two domains. It is scored using a 6-point Likert scale and has been validated in Brazilian Portuguese, French, Spanish, and Japanese .Therefore, the aim of this study was to adapt the KNAP questionnaire for Turkish physiotherapists and to rigorously examine its psychometric properties among physiotherapy graduates and students in Turkey. The study aims to validate the questionnaire to accurately assess pain knowledge, attitudes, and beliefs by analyzing internal consistency, structural and construct validity, reliability, sensitivity, and interpretability.

ELIGIBILITY:
Inclusion Criteria: Physiotherapy and rehabilitation department students and physiotherapists who speak Turkish -

Exclusion Criteria: Physiotherapy and rehabilitation students and physiotherapists who do not speak Turkish.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physiotherapy and rehabilitation department students and physiotherapists who speak Turkish
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-05 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
KNAP | 10 minutes
  The Knowledge and Attitudes of Pain (KNAP) questionnaire was developed to address these limitations, evaluating the knowledge of modern pain science and biopsychosocial attitudes toward pain

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gokhan MARAS, Ankara
  - Gökhan maraş, Ankara

IPD SHARING:
Plan to Share IPD: Undecided